CLINICAL TRIAL: NCT05719532
Title: Correlation of Core Strength/Core Stability and Coordinative Skills in Healthy Adults - an Explorative Study
Brief Title: Core Strength and Coordinative Skills
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Johannes Kepler University of Linz (Other)
Collaborators: Kepler University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PMR_Core_Balance_001
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Postural Balance; Core Strength; Core Stability; Physical Fitness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy adults: Healthy adults between 18 and 35 years

SUMMARY:
Evaluation of healthy young adults regarding balance, core strength/core stability and physical fitness. Correlation of primary outcome parameters and selected secondary parameters.

ELIGIBILITY:
Inclusion Criteria:

* Adequat cognitive and lingual competence
* Written informed consent

Exclusion Criteria:

* low back pain or other painful disorders regarding the spine during the last 6 weeks
* Previous spine surgery
* Neurologic disease or disease of the vestibular organ
* Previous arthroplasty of joints

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy young adults between 18 and 35 years.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-03-29 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Center of pressure track (COPT) | Baseline
  Posturographic parameter; lower values indicate better postural stability
Area of sway (AOS) | Baseline
  Posturographic parameter; lower values indicate better postural stability
Core stability test of the Swiss Olympic Medical Center | Baseline
  Measurement of Core strength/Core stability in sec; higher values indicate better core strength

SECONDARY OUTCOMES:
Baecke Questionnaire of Habitual Physical Activity (BQHPA) | Baseline
  Questionnaire of physical fitness; higher values indicate higher physical fitness
Stability energy | Baseline
  Posturographic parameter, measures economy of movement; higher values mean lower stabilty
Harmony index | Baseline
  Posturographic parameter
Frequency of sway | Baseline
  Posturographic parameter
Feedback | Baseline
  Posturographic parameter; quantitative data; a score is calculated by the posturographic system to determine the influence of visual, vestibular and somatosensory feedback on postural control
Movement control | Baseline
  Posturographic parameter; the frequencies of the movement amplitude during the posturographic measurement are calculated and a score for the low and high frequencies is presented. For the lower frequencies (F1, F2) higher values are positive. For the higher frequencies (F3 - F8) lower values are positive.
Weight distribution index | Baseline
  Posturographic parameter; Center of pressure at beginning of measurement
Body mass index (BMI) | Baseline
  Relation weight to height

CONTACTS AND LOCATIONS:
Overall Officials: Christian Mittermaier, M.D., Principal Investigator — Kepler University Hospital
Locations (1):
- Department of Physical Medicine & Rehabilitation, Kepler University Hospital, Linz, Austria